CLINICAL TRIAL: NCT04027088
Title: Multicenter Randomized Clinical Trial of the Effect of Preoperative Immunonutrition Versus Standard Enteral Nutrition in Elective Oncological Surgery of the Upper Digestive Tract
Brief Title: Effect of Preoperative Immunonutrition in Upper Digestive Tract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Alfonso Vidal Casariego, Dr. Alfonso Vidal Casariego, MD PhD, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2018/548
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Immunonutrition; Gastric Cancer; Esophageal Cancer; Pancreas Cancer; Surgery--Complications
Keywords: immunonutrition; surgery; postoperative complications; length of hospital stay; nutritional status
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition (Experimental): Oral nutritional supplement: hypercaloric and hyperproteic with immunonutrients: Arginine, nucleotides, omega-3, olive oil polyphenols, antioxidants and L-carnitine
  Interventions: Dietary Supplement: Immunonutrition
- Standard (Placebo Comparator): Oral nutritional supplement: hypercaloric and hyperproteic without immunonutrients
  Interventions: Dietary Supplement: Standard

INTERVENTIONS:
Dietary Supplement: Immunonutrition — It is a hypercaloric and hyperproteic dietary supplement formulated with immunonutrients: Arginin, nucleotides, omega-3, olive oil polyphenols, antioxidants and L-carnitine
  Other Names: Bi1 procare
  Arms: Immunonutrition
Dietary Supplement: Standard — It is a hypercaloric and hyperproteic dietary supplement formulated without immunonutrients
  Arms: Standard

SUMMARY:
Randomized, double-blind, multicenter clinical trial that will evaluate the effects of immuno-nutrition in the preoperative period in patients with cancer of the upper digestive tract (esophagus, stomach, and pancreas). The aim is to compare the specific effect of the immunonutrients respect to an equivalent formula in caloric-protein value but without immunonutrients, in the surgical evolution of the cancer patient.

DETAILED DESCRIPTION:
Background:

Perioperative nutritional status is a key factor in the evolution, as well as, postoperative morbidity and mortality of cancer patients. Particularly, digestive neoplasms have a high risk of malnutrition and this is related to a higher rate of surgery complications and mortality in the postoperative period. The immunonutrition seems to modulate the immune system and the inflammatory response in patients operated on for digestive neoplasia. However, the results to date are controversial.

Aim:

To compare the effect of an immunomodulatory oral nutritional supplement (enriched in arginine, nucleotides, omega 3 fatty acids, olive oil polyphenols, L-carnitine, and antioxidants) against an equivalent in protein-energy without immunonutrients, administrated in the preoperative period, in the surgical evolution of the cancer patient with neoplasia of the upper digestive tract.

Methods:

It is a randomized, double-blind, multicenter clinical trial. 178 patients with neoplasms of the esophagus, stomach or pancreas, with indication of surgical treatment, will be included. The patients will be randomized into two groups (intervention group and control group) and both will receive 2 daily bricks of the assigned formula (with or without immunonutrients, respectively) 5 days prior to surgery. The main variables of the study are: appearance of infectious or noninfectious complications in the postoperative period, length of hospital stay, and mortality. These variables will be compared by group (immunonutrition vs. non immunonutrition).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer of esophagus, stomach and / or pancreas, at any stage, proposed for surgery
* Signing informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Advanced renal insufficiency prior to dialysis (GFR <25 ml / min)
* Allergy or intolerance to any of the components of the dietary supplement (including fish allergy)
* Patients with contraindications for enteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Infectious complications | Up to 30 days post-operative
Surgical fistulas | Up to 30 days post-operative

SECONDARY OUTCOMES:
Mortality | Up to 30 days post-operative
Length of hospital stay | Up to 30 days post-operative
Weight loss | 10 days Pre-operative

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Á Martínez-Olmos, PhD, MD, Principal Investigator — Complexo Hospitalario Universitario de Santiago; Alfonso Vidal-Casariego, PhD, MD, Principal Investigator — Complexo Hospitalario Universitario de A Coruña
Locations (2):
- Spain (2):
  - Miguel A. Martínez Olmos, Santiago de Compostela, A Coruña
  - Alfonso Vidal-Casariego, A Coruña, La Coruna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villar-Taibo R, Vidal-Casariego A, Santamaria-Nieto A, Canton-Blanco A, Crujeiras AB, Lugo Rodriguez G, Rodriguez-Carnero G, Pita Gutierrez F, Fernandez Pombo A, Diaz-Lopez E, Roman Eyo A, Rodriguez Lavandeira U, Pena-Dubra A, Martinez-Olmos MA. Efficacy of a new immunonutrition formula with extra virgin olive oil in the reduction of complications in surgeries of upper digestive tract tumors. Front Nutr. 2024 May 28;11:1384145. doi: 10.3389/fnut.2024.1384145. eCollection 2024. PMID 38863591